CLINICAL TRIAL: NCT07268664
Title: Innovating Shorter, All- Oral, Precised Treatment Regimen for Rifampicin Resistant Tuberculosis：BLMZ Chinese Cohort
Acronym: INSPIRE-BLMZ
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Chest Hospital (Other)
Collaborators: National Medical Center for Infectious Diseases (Unknown); Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chu naihui, Professor, Beijing Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJCH-202509
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Rifampicin Resistant Tuberculosis; Pulmonary Tuberculosis; Tuberculosis; Drug-resistant Tuberculosis
Keywords: drug-resistant tuberculosis; all-oral regimen; 9 month regimen; tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis; Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): All enrolled participants will receive the all-oral, shorter-course BLMZ regimen for a total of 9 months from end-TB study, as described in the Intervention section.
  Interventions: Drug: BLMZ

INTERVENTIONS:
Drug: BLMZ — The regimen is composed of the following four drugs, with doses adjusted by body weight:
  Bedaquiline (BDQ):
  * Weeks 1-2: 400 mg (two 200 mg tablets) orally, once daily.
  * Weeks 3 to Month 9: 200 mg orally, three times per week (with at least 48 hours between doses).
  Linezolid (LZD):
  * Months 1-4: 600 mg orally, once daily.
  * Months 5-9: Dose reduced to 300 mg orally, once daily (or an intermittent dosing strategy) for the remainder of treatment. Earlier dose adjustment is permitted in cases of drug intolerance or related adverse events.
  Moxifloxacin (MFX):
  - 400 mg orally, once daily throughout the 9-month treatment.
  Pyrazinamide (PZA):
  - Administered orally, once daily at a weight-based dose: 750 mg for participants weighing 30-34.9 kg 1000 mg for participants weighing 35-49.9 kg 1500 mg for participants weighing ≥50 kg

SUMMARY:
The goal of this clinical trial is to learn if the all-oral, shorter-course BLMZ regimen can treat Rifampicin-Resistant Tuberculosis (RR-TB) in Chinese participants aged 12 years and older. The main questions it aims to answer are:

What is the proportion of participants with a favorable outcome at 18 months after starting the BLMZ regimen? What is the safety profile of the BLMZ regimen, as measured by the incidence of Grade 3 or higher adverse events and serious adverse events during the treatment period? This is a single-arm study, so there is no comparison group. Researchers will compare the study results to historical data to see if the BLMZ regimen shows sufficient efficacy and safety in the Chinese population.

Participants will:

Undergo screening tests to confirm eligibility, including tests for TB bacteria and drug resistance.

Receive the BLMZ regimen (Bedaquiline, Linezolid, Moxifloxacin/Levofloxacin, and Pyrazinamide) orally for 9 months.

Attend regular clinic visits for safety assessments, medication refills, and tests (e.g., sputum tests, blood tests, ECG, CT scans) during the 9-month treatment period and then every 3 months during a 15-month post-treatment follow-up period until 24 months after starting the treatment.

DETAILED DESCRIPTION:
Study Rationale and Background:

Tuberculosis (TB) remains a significant global health threat, with Rifampicin-Resistant TB (RR-TB) posing a particularly severe challenge due to prolonged treatment durations, high toxicity, and suboptimal success rates. While the standard of care in China has historically involved 18-20 month regimens, the World Health Organization (WHO) has recently endorsed shorter, all-oral regimens. The BLMZ regimen, composed of Bedaquiline (B), Linezolid (L), Moxifloxacin (M), and Pyrazinamide (Z), demonstrated high efficacy (89% favorable outcome) in the global endTB trial. However, prospective data on its application and performance in the Chinese population are lacking. This study aims to bridge this evidence gap by prospectively evaluating the efficacy, safety, and feasibility of the 9-month BLMZ regimen in a Chinese RR-TB cohort, thereby informing national policy and clinical practice.

Study Design:

This is a prospective, multicenter, single-arm, open-label, interventional study. The study employs a Bayesian statistical framework with a pre-specified success threshold to evaluate the primary efficacy endpoint. Historical data from the endTB study (BLMZ arm) will be incorporated using a power prior model to augment the statistical analysis, allowing for more robust inference with the planned sample size.

Intervention:

Participants will receive the all-oral BLMZ regimen for a total of 9 months. The regimen consists of:

* Bedaquiline (BDQ): 400 mg once daily for 2 weeks, followed by 200 mg three times per week for the remainder of the 9-month treatment.
* Linezolid (LZD): 600 mg once daily for the first 4 months, followed by a dose reduction to 300 mg once daily (or intermittent dosing) for the remaining 5 months, with provisions for earlier adjustment in case of intolerance.
* Moxifloxacin (MFX): 400 mg once daily. In cases of MFX unavailability, intolerance, or resistance, it may be substituted with Levofloxacin (LFX) at a weight-based dose (750 mg for 35-49.9 kg, 1000 mg for ≥50 kg).
* Pyrazinamide (PZA): Administered at a weight-based dose (750 mg for 30-34.9 kg, 1000 mg for 35-49.9 kg, 1500 mg for ≥50 kg) once daily.

Drug doses are adjusted according to pre-specified weight bands. Treatment may be extended to a maximum of 11 months under specific conditions (e.g., positive culture at Month 2, unclosed cavity at Month 9).

Study Population and Follow-up:

The study will enroll approximately 120 participants aged ≥12 years with bacteriologically confirmed pulmonary RR-TB who are susceptible to fluoroquinolones. Participants may be either treatment-naïve or previously treated for drug-susceptible TB.

The study duration for each participant is 24 months, comprising:

Screening Period: Up to 4 weeks. Treatment Period: 9 months (extendable to 11 months), with monthly on-site visits for clinical, bacteriological (sputum smear and culture), and safety assessments (including hematology, biochemistry, electrolytes, visual acuity, peripheral neuropathy screening, and 12-lead ECG). Chest CT scans are performed at baseline, Month 5, and Month 8.

Post-Treatment Follow-up Period: 15 months, with quarterly visits until Month 24. Follow-up focuses on long-term efficacy and safety, primarily through sputum culture for relapse detection.

Key Technical and Operational Considerations:

1. Outcome Definitions: Favorable and unfavorable outcomes at 9, 18, and 24 months are rigorously defined based on a composite of bacteriological results, treatment modifications, and clinical status, aligning with contemporary TB trial standards.
2. Safety Monitoring: A comprehensive safety management plan is in place. Special attention is given to Adverse Events of Special Interest (AESI), including hepatotoxicity, QT interval prolongation, optic neuropathy, and peripheral neuropathy, with predefined grading and reporting procedures.
3. Concomitant Medication Restrictions: The protocol explicitly prohibits the use of strong CYP3A4 inducers/inhibitors, monoamine oxidase inhibitors, drugs known to cause significant QT prolongation or bone marrow suppression, to minimize drug-drug interactions and overlapping toxicities.
4. Management of Non-Adherence and Interruptions: The protocol allows for temporary treatment interruptions and defines criteria for permanent discontinuation. Strategies to promote adherence are implemented, and the impact of interruptions on the overall treatment duration is clearly specified.
5. Statistical Analysis Plan: The primary analysis will be conducted on the modified Intent-to-Treat (mITT) population. The Bayesian decision rule for success is defined as a posterior probability >0.95 that the true favorable outcome rate at 18 months is ≥85%. A simulation study was conducted to determine the optimal sample size (n=120) and the power prior weight (ω=0.35) to control Type I error and ensure adequate statistical power.
6. Quality Assurance: The study will be conducted under the principles of Good Clinical Practice (GCP). Data quality will be ensured through centralized monitoring, risk-based source data verification, and regular site training and oversight.

ELIGIBILITY:
Inclusion Criteria:

* The participant (and their guardian if the participant lacks civil capacity) voluntarily signs the informed consent form (ICF) prior to enrollment.
* The participant (and their guardian) indicates willingness to complete all steps and intervention periods of the study.
* Male or female, aged ≥12 years, with a body weight ≥30 kilograms (kg).
* Bacteriologically confirmed pulmonary tuberculosis, with molecular or phenotypic drug susceptibility testing (DST) results within the last 3 months confirming Rifampicin resistance and susceptibility to at least one of Moxifloxacin (MFX) or Levofloxacin (LFX).
* Sputum or respiratory lavage fluid collected during the screening period is culture-positive for Mycobacterium tuberculosis, with DST results indicating Rifampicin resistance and susceptibility to at least one of MFX or LFX.
* Females of childbearing potential are not pregnant (as confirmed by a negative pregnancy test), voluntarily agree to pregnancy testing, and are willing to use highly effective contraception from the time of ICF signing until 3 months after the end of study treatment.
* For males of reproductive potential, use condoms or other methods to ensure effective contraception for their partner.
* Females who are breastfeeding are willing to discontinue breastfeeding from the time of ICF signing until 3 months after the end of study treatment.
* Voluntary acceptance of HIV testing; if the result is positive, voluntary acceptance of antiretroviral therapy.

Exclusion Criteria:

* Previous treatment with any of the drugs Bedaquiline (BDQ) or Linezolid (LZD) for more than 30 days.
* Concurrent hematogenous disseminated pulmonary tuberculosis or severe extrapulmonary tuberculosis as determined by the investigator.
* Current use of medications prohibited by the study protocol, and the investigator judges that the priority of continuing said medication for patient benefit outweighs participation in this study.

（Note: If the investigator judges that the benefit of participating in this study is higher and obtains the participant's consent, the prohibited medication should be discontinued with an adequate washout period before participation.）

* Known history of hypersensitivity to any drug in the protocol.
* Current participation in any other investigational drug clinical trial.
* Presence of cardiovascular disease risk at screening:

  1. QTcF interval >450 milliseconds (ms). (Note: If QTcF >450 ms is detected, one unscheduled visit during the screening period is allowed for re-assessment.)
  2. History of clinically significant arrhythmia within 60 days prior to enrollment, which in the investigator's opinion may increase risk upon study participation.
  3. Decompensated heart failure.
  4. Grade 3 hypertension not at control target.
  5. Abnormal thyroid function.
  6. Abnormal serum calcium, magnesium, or potassium levels. (Note: Isolated electrolyte disturbances without underlying disease may be considered for re-screening after corrective treatment.)
  7. Other conditions deemed by the investigator to pose a cardiovascular disease risk.
* History of optic neuropathy or peripheral neuropathy, which in the investigator's opinion may progress/worsen during the study or is unsuitable for study participation.
* Evidence of liver disease at screening:

  1. Active viral hepatitis: Positive HBsAg, or positive HBeAg and HBV DNA, or positive HCV RNA test, accompanied by persistent or recurrent abnormal ALT.
  2. Decompensated cirrhosis.
* History of renal disease or renal disease-related manifestations at screening:

  1. History of unstable or rapidly progressive renal disease.
  2. Moderate/severe renal impairment or end-stage renal disease (eGFR < 60 mL/min/1.73 m²).
  3. Serum creatinine (Cr) ≥133 μmol/L (1.5 mg/dL) for males, or Cr ≥124 μmol/L (1.4 mg/dL) for females.
* Other laboratory abnormalities at screening:

  1. Hemoglobin level < 8.0 g/dL.
  2. Platelet count <75,000 /mm³.
  3. Absolute neutrophil count (ANC) <1000 /mm³.
  4. Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) >3 times the upper limit of normal (ULN).
  5. Total bilirubin >2 times ULN, or >1.5 times ULN accompanied by other abnormal liver enzymes.
  6. Albumin <30 g/L.
* Pregnant or breastfeeding.
* Any other condition (e.g., severe psychiatric disorder, neurological condition, substance abuse) that, in the opinion of the investigator, would make the participant unsuitable for the study or unable to adhere to the protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with favorable outcome | 18 months after treatment initiation
  Favorable Outcome: A participant is considered to have a favorable outcome if they do not meet any criteria for an unfavorable outcome, and they meet the following key criterion: two consecutive negative sputum cultures, with the final culture obtained between 16 and 18 months after treatment initiation.
  Unfavorable Outcome: An outcome is classified as unfavorable if any of the following occur:
  * Treatment failure (change of regimen).
  * Extended treatment beyond the protocol-defined period.
  * Bacteriological relapse or failure (positive culture at the end of the study period).
  * Death from any cause.
  * Loss to follow-up.

SECONDARY OUTCOMES:
The proportion of participants with favorable outcome | 9 months after treatment initiation
The proportion of participants with favorable outcome | 24 months after treatment initiation
The proportion of participants with sputum conversion | 2 months from treatment initiation
Time to sputum conversion | 9 months after treatment initiation
the incidence of grade 3 or worse AEs and SAEs | 24 months after treatment initiation
  As measured by

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Third People's Hospital in Aksou, Aksu, Xinjiang
  - Hetian Prefecture Infectious Diseases Hospital, Hetian, Xinjiang
  - Center of Disease Prevention and Control in Kashi Area, Kashgar, Xinjiang

IPD SHARING:
Plan to Share IPD: Yes